CLINICAL TRIAL: NCT04909320
Title: Building Capacity and Promoting Smoking Cessation in the Community Via "Quit to Win" Contest 2021: Mobile-based Positive Psychological Support on Smoking Cessation
Brief Title: Mobile-based Positive Psychological Support for Smoking Cessation Via "Quit to Win" Contest 2021 (QTW 2021)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Council on Smoking and Health (Other)
Responsible Party: Principal Investigator, Dr. Wang Man-Ping, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: QTW 2021
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Smoking Cessation
Keywords: smoking cessation; positive psychological support; mobile health; peer supporter
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Behavioral: AWARD advice; Other: Brief leaflet on health warning and smoking cessation; Other: Referral card; Other: Self-help smoking cessation booklet; Behavioral: Positive psychological support through 3-people group chat using instant messaging apps
- Control group (Active Comparator)
  Interventions: Behavioral: AWARD advice; Other: Brief leaflet on health warning and smoking cessation; Other: Referral card; Other: Self-help smoking cessation booklet; Behavioral: E-messages via SMS

INTERVENTIONS:
Behavioral: AWARD advice — Ask about smoking history; Warn about the high risk; Advise to quit; Refer smokers to smoking cessation services (with a referral card); Do it again
Other: Brief leaflet on health warning and smoking cessation — The contents of the leaflet include (1) highlights of the absolute risk of death due to smoking; (2) the whole list of diseases caused by active and second-hand smoking; (3) ten horrible pictorial warnings of health consequences of smoking and second-hand smoking in one page to maximize the impacts; (4) benefits of SC and (5) simple messages to encourage participants to quit smoking and remind them to call the Department of Health SC hotline 183 3183.
Other: Referral card — The contents consist of brief information and highlights of existing SC services, contact methods, motivation information, and strong supporting messages or slogans.
Other: Self-help smoking cessation booklet — The contents include information about the benefits of quitting, smoking and diseases, methods to quit, how to handle withdrawal symptoms, declaration of quitting, etc.
Behavioral: Positive psychological support through 3-people group chat using instant messaging apps — Each IM chat group will consist of a trained SC counselor (HKU staff), a peer supporter (former smoker), and a participant (smoker). The 3-month group chat-based intervention will consist of regular messages and real-time support through group chat. Regular messages will generally include goal setting, health warnings, abstinence support, positive psychological exercises, and encouragement and will be delivered in a tapering style. During the real-time chatting, SC counsellors and peer supporters will provide real-time chat-based support, and peer supporters will share their quitting experience as appropriate.
  Arms: Intervention group
Behavioral: E-messages via SMS — Regular e-messages via SMS at twice per month within 3 months (total 6).
  Arms: Control group

SUMMARY:
This study aims to explore the effectiveness of a combined intervention using brief cessation advice and personalized chat-based positive psychological support compared with the control group on current smokers who join the Quit to Win Contest.

DETAILED DESCRIPTION:
Smoking is a leading cause of many diseases and deaths globally. Although Hong Kong has a relatively low overall smoking rate of 10.2% (in 2019), health and economic burdens due to smoking are still substantial. The practice of smoking might predispose smokers to COVID-19 infection and poor prognosis. Growing evidence has also suggested that smokers are at higher risk of developing serious respiratory and cardiovascular symptoms in the COVID-19 pandemic than non-smokers. Smoking cessation in the post-COVID-19 era is the key priority to meet the HKSAR Government's target of reducing smoking prevalence to 7.8% by 2025.

Mental health problems are commonly comorbid with smoking and related problems. Our population-based survey amidst the COVID-19 pandemic found current smokers were at higher risk of suffering from anxious symptoms (adjusted OR 1.84 95% CI 1.27, 2.67), depressive symptoms (adjusted OR 2.04 95% CI 1.40, 2.96), and stress symptoms (adjusted β 0.54 95% CI 0.26, 0.82) compared with non-smokers. We also observed mental health burden increased during the COVID-19 pandemic with approximately doubling of the prevalence of anxious symptoms (15.8 vs. 9.3) and depressive symptoms (14.8 vs. 6.3) compared with the pre-COVID-19 pandemic (2017). Mental health can be both precursors and consequences of smoking. Previous studies have suggested that depressive symptoms and low positive affect during and after SC attempts are associated with poor cessation outcomes. This implies that a combined intervention of behavioral and psychological SC intervention is needed, particularly under the circumstance of worsening mental health problems.

Therefore, our study aims to test the effectiveness of a combined intervention using brief cessation advice and personalized chat-based positive psychological support compared with the control group on current smokers who join the Quit to Win Contest.

ELIGIBILITY:
Inclusion Criteria:

* Hong Kong residents aged 18 or above
* Smoke at least 1 tobacco stick (includes HTP) per day or use e-cigarette daily in the past 3-month
* Able to communicate in Chinese
* Saliva cotinine 30 ng/ml or above
* Intent to quit/reduce smoking
* Able to use the instant messaging tool (e.g., WhatsApp, WeChat) for communication

Exclusion Criteria:

* Smokers who have communication barrier (either physically or cognitively)
* Smokers who are currently participating in other SC programmes or services

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1094 (Estimated)
Dates: Start 2021-06-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Biochemically validated abstinence | 6-month follow-up
  Defined as exhaled CO level <4ppm and saliva cotinine level ≤30 ng/ml
  Note
  1. If participants refuse to have a face-to-face exhaled carbon monoxide test due to the COVID-19 pandemic in Hong Kong. In that case, the outcome will only be validated by a saliva cotinine test device.
  2. If participants use NRT, the outcome will be validated by exhaled carbon monoxide only.

SECONDARY OUTCOMES:
Biochemically validated abstinence | 3-month follow-up
  Defined as exhaled CO level <4ppm and saliva cotinine level ≤30 ng/ml
  Note
  1. If participants refuse to have a face-to-face exhaled carbon monoxide test due to the COVID-19 pandemic in Hong Kong. In that case, the outcome will only be validated by a saliva cotinine test device.
  2. If participants use NRT, the outcome will be validated by exhaled carbon monoxide only.
Self-reported 7-day point prevalence quit rate | 3-month follow-up
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up
Self-reported 7-day point prevalence quit rate | 6-month follow-up
  Smokers who did not smoke even a puff in the 7 days preceding the follow-up
Self-reported reduction | 3-month follow-up
  Defined by at least 50% reduction in baseline daily number of cigarettes
Self-reported reduction | 6-month follow-up
  Defined by at least 50% reduction in baseline daily number of cigarettes
Self-reported depressive symptoms | 3-month follow-up
  Measured by Patient Health Questionnaire-2 (PHQ-2). PHQ-2 ranges from 0-6, a higher score indicates a severer depressive symptom.
Self-reported depressive symptoms | 6-month follow-up
  Measured by Patient Health Questionnaire-2 (PHQ-2). PHQ-2 ranges from 0-6, a higher score indicates a severer depressive symptom.
Self-reported anxious symptoms | 6-month follow-up
  Measured by Generalized Anxiety Disorder-2 (GAD-2). GAD-2 ranges from 0-6, a higher score indicates a severer anxious symptom.
Self-reported anxious symptoms | 3-month follow-up
  Measured by Generalized Anxiety Disorder-2 (GAD-2). GAD-2 ranges from 0-6, a higher score indicates a severer anxious symptom.
Self-reported use of smoking cessation service | 3-month follow-up
  Use of smoking cessation service at 3- and 6- month follow-up
Self-reported use of smoking cessation service | 6-month follow-up
  Use of smoking cessation service at 3- and 6- month follow-up
Self-rated health | 3-month follow-up
  Self-rated health will be measured as a single item with the response items "excellent", "very good", "good", "fair", or "poor".
Self-rated health | 6-month follow-up
  Self-rated health will be measured as a single item with the response items "excellent", "very good", "good", "fair", or "poor".
Self-reported happiness | 3-month follow-up
  A single item will measure self-reported happiness with an answer on an 11-point scale (0-10). A higher score indicates a higher level of happiness.
Self-reported happiness | 6-month follow-up
  A single item will measure self-reported happiness with an answer on an 11-point scale (0-10). A higher score indicates a higher level of happiness.
Self-reported quit attempts | 3-month follow-up
  Number of quit attempts from baseline at 3-month follow-up
Self-reported quit attempts | 6-month follow-up
  Number of quit attempts from baseline at 6-month follow-up
Self-reported resilience | 3-month follow-up
  A single item will measure self-reported resilience with an answer on an 11-point scale (0-10). A higher score indicates a higher level of resilience.
Self-reported resilience | 6-month follow-up
  A single item will measure self-reported resilience with an answer on an 11-point scale (0-10). A higher score indicates a higher level of resilience.
Self-reported optimistic | 3-month follow-up
  A single item will measure self-reported optimistic with an answer on an 11-point scale (0-10). A higher score indicates a higher level of optimistic.
Self-reported optimistic | 6-month follow-up
  A single item will measure self-reported optimistic with an answer on an 11-point scale (0-10). A higher score indicates a higher level of optimistic.
Self-reported loneliness | 3-month follow-up
  A single item will measure self-reported loneliness with an answer on an 11-point scale (0-10). A higher score indicates a higher level of loneliness.
Self-reported loneliness | 6-month follow-up
  A single item will measure self-reported loneliness with an answer on an 11-point scale (0-10). A higher score indicates a higher level of loneliness.
Self-reported stress | 6-month follow-up
  A single item will measure self-reported stress with an answer on an 11-point scale (0-10). A higher score indicates a higher level of stress.
Self-reported stress | 3-month follow-up
  A single item will measure self-reported stress with an answer on an 11-point scale (0-10). A higher score indicates a higher level of stress.
Self-reported social support | 3-month follow-up
  A single item will measure self-reported social support with an answer on an 11-point scale (0-10). A higher score indicates a higher level of social support.
Self-reported social support | 6-month follow-up
  A single item will measure self-reported social support with an answer on an 11-point scale (0-10). A higher score indicates a higher level of social support.
Self-reported positive affect | 3-month follow-up
  The subscale of the Chinese version International Positive and Negative Affect Schedule Short Form (I-PANAS-SF) will measure self-reported positive affect. The I-PANAS-SF uses a 5-point scale, a higher score indicates a higher level of self-reported positive affect.
Self-reported positive affect | 6-month follow-up
  The subscale of the Chinese version International Positive and Negative Affect Schedule Short Form (I-PANAS-SF) will measure self-reported positive affect. The I-PANAS-SF uses a 5-point scale, a higher score indicates a higher level of self-reported positive affect.
Self-reported negative affect | 6-month follow-up
  The subscale of the Chinese version International Positive and Negative Affect Schedule Short Form (I-PANAS-SF) will measure self-reported negative affect. The I-PANAS-SF uses a 5-point scale, a higher score indicates a higher level of self-reported negative affect.
Self-reported negative affect | 3-month follow-up
  The subscale of the Chinese version International Positive and Negative Affect Schedule Short Form (I-PANAS-SF) will measure self-reported negative affect. The I-PANAS-SF uses a 5-point scale, a higher score indicates a higher level of self-reported negative affect.

CONTACTS AND LOCATIONS:
Overall Officials: Man Ping Wang, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Hong Kong Council on Smoking and Health (COSH), Hong Kong, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo Z, Luk TT, Weng X, Wu Y, Zhao S, Lai YK, Cheung DYT, Tong HSC, Lai VWY, Lam TH, Wang MP. Behavioral Support by Ex-Smoking Peers Using Instant Messaging for Smoking Cessation: A Randomized Controlled Trial. Chest. 2026 Jan;169(1):300-311. doi: 10.1016/j.chest.2025.07.4110. Epub 2025 Sep 10. PMID 40939935